CLINICAL TRIAL: NCT01828502
Title: Cotinine Feedback as an Intervention to Change Parental/Caregiver Smoking Behavior Around Children With Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed due to poor accrual. No patients were enrolled.
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SCUSF 1201
Record Dates: First submitted 2013-03-28; First posted 2013-04-10 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Pediatric Cancer
Keywords: Cotinine; Secondhand Smoke Exposure (SHSE); Secondhand Smoke (SHS)
MeSH Terms: conditions — Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Intervention (Experimental): Those randomized to the active intervention will receive education about secondhand smoke exposure and feedback using the cotinine test strip.
  Interventions: Behavioral: Education; Behavioral: Cotinine Education
- Education only (Other): Those randomized to the education only group will receive only the education about secondhand smoke exposure.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Participants in both groups will receive education by the EPA on the danger of exposure to secondhand smoke and how exposure can be prevented.
Behavioral: Cotinine Education — Those randomized to the active intervention will also be provided with education utilizing the cotinine test strip in conjunction with the education from the EPA.
  Arms: Active Intervention

SUMMARY:
RATIONALE: Providing parent/caregivers of children with cancer with education and evidence of secondhand smoke exposure can protect the child from future exposure to tobacco smoke.

PURPOSE: This randomized study will compare education only to education plus cotinine feedback in decreasing secondhand smoke exposure in pediatric patients with cancer that reside with a household smoker.

DETAILED DESCRIPTION:
OBJECTIVES:

The primary objective of this study is to determine if providing urine cotinine feedback to caregivers in conjunction with standard education will be more effective than education alone in reducing patient SHS exposure.

The secondary objectives of this study are:

To determine whether urine cotinine feedback in conjunction with education provided to the caregiver is more effective in changing parental smoking behavior compared to education alone.

As an exploratory measure we will collect history and physical exam data to follow patient's clinical complications during the study to determine if patients with a decrease in SHS exposure also have a decrease in clinical complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 years and ≤ 12 years at the time of study entry.
* Currently undergoing treatment for cancer at the time of enrollment, at least 28 days post diagnosis.
* The child must reside 5 days a week with a household smoker (defined as a person who smokes greater than 10 cigarettes daily).
* Child must be potty trained.
* Parent/Legal Guardian ≥ 18 years of age.
* Parent/Legal Guardian who accompanies the child to the first visit must accompany the child to all other visits. This person does not need to be the household smoker, but must be willing to educate the smoker on results at the visit and take the education handout home to them.
* Parent/Legal Guardian must have a working phone to complete the week 5 follow-up phone call.
* Able and willing to sign informed consent/assent.
* Signed HIPAA compliant research authorization.

Exclusion Criteria:

* Planned hospitalization within 3 days of any scheduled study visit (due to the urine cotinine measurement representing the previous 48-72 hours of tobacco exposure.
* Inability to perform the initial cotinine test.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in urine cotinine level | 4 weeks after baseline visit
  The primary objective of this study is to determine if providing urine cotinine feedback to caregivers in conjunction with standard education will be more effective than education alone in reducing patient SHS exposure.

SECONDARY OUTCOMES:
Change in Self-Reported Smoking Behavior | 4 weeks after baseline visit
  To determine whether urine cotinine feedback in conjunction with education provided to the caregiver is more effective in changing parental smoking behavior compared to education alone.
Number of medical complications | 4 weeks after baseline visit
  As an exploratory measure we will collect history and physical exam data to follow patient's clinical complications during the study to determine if patients with a decrease in SHS exposure also have a decrease in clinical complications.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Couluris, DO, Study Chair — University of South Florida
Locations (10):
- United States (10):
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lee Memorial Hospital - The Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic, Pensacola, Florida
  - All Children's Hospital, Saint Petersburgh, Florida
  - Tampa General Hospital, Tampa, Florida
  - Columbia University Medical Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - St. Vincent Hospital, Green Bay, Wisconsin